CLINICAL TRIAL: NCT00883558
Title: A Phase II, Randomized, Open Label, 2-Way Crossover, Safety Study of Subcutaneously Injected Prandial INSULIN-PH20 NP Compared to Insulin Analog Injection in Patients With Type 1 Diabetes
Brief Title: Safety Study of Subcutaneously-Injected Prandial INSULIN-PH20 NP Compared to Insulin Lispro Injection in Participants With Type 1 Diabetes Mellitus
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Halozyme Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: HALO-117-203
Record Dates: First submitted 2009-04-15; First posted 2009-04-17 (Estimated); Results first posted 2014-09-08 (Estimated); Last update posted 2014-09-08 (Estimated); Status verified 2014-08

CONDITIONS: Diabetes Mellitus, Type 1
Keywords: recombinant human hyaluronidase (rHuPH20); Insulin lispro; regular human insulin
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Insulin Resistance | interventions — Insulin Lispro; Insulin; Insulin Glargine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- INSULIN-PH20 NP / Insulin Lispro (Experimental): All enrolled participants underwent a 1-month dose titration period and received 100 units per milliliter (U/mL) insulin lispro, injected subcutaneously (SC) pre-meals, with doses titrated to each participant individually.
  Next participants were randomly assigned to 1 of 2 study treatments (Treatment A or B) for the first of two, 3-month treatment cycles. Each participant then received the second treatment for the second cycle.
  INSULIN-PH20 NP (Treatment A): 100 U/mL non-preserved (NP) formulation of regular human insulin with 5.0 micrograms per milliliter (µg/mL) recombinant human hyaluronidase PH20, injected SC, pre-meals, doses titrated to each participant individually.
  Insulin Lispro (Treatment B): 100 U/mL insulin lispro, injected SC, pre-meals, doses titrated to each participant individually.
  Throughout the study, participants requiring basal insulin used twice daily SC injections of 100 U/mL insulin glargine or maintained their usual regimen through an insulin pump.
  Interventions: Drug: Insulin Lispro; Drug: regular human insulin; Drug: recombinant human hyaluronidase PH20; Drug: Insulin glargine

INTERVENTIONS:
Drug: Insulin Lispro
  Other Names: Humalog
Drug: regular human insulin
  Other Names: Humulin R
Drug: recombinant human hyaluronidase PH20
  Other Names: Hylenex; rHuPH20; PH20
Drug: Insulin glargine
  Other Names: Lantus

SUMMARY:
Insulin lispro is approved by the Food and Drug Administration (FDA) for the treatment of diabetes mellitus. Recombinant human hyaluronidase (rHuPH20) is approved by the FDA as an aid to the absorption and dispersion of other injectable drugs. In this study, rHuPH20 combined with a non-preserved (NP) formulation of regular human insulin (INSULIN-PH20 NP) will be compared to insulin lispro with respect to absorption and action of insulin.

DETAILED DESCRIPTION:
The purpose of this study is to compare the safety and tolerability of INSULIN-PH20 NP versus insulin lispro alone.

ELIGIBILITY:
Inclusion Criteria:

* Male or female of age 18 to 65 years, inclusive. Females of child-bearing potential must use a standard and effective means of birth control for the duration of the study.
* Participants with Type 1 diabetes mellitus (T1DM) (per World Health Organization [WHO] criteria) treated with insulin for ≥24 months.
* Participants who use an insulin infusion pump for basal insulin administration must be on the device for at least 90 days prior to screening.
* Body mass index (BMI) 18.0 to 35.0 kilograms per square meter (kg/m^2), inclusive.
* Glycosylated hemoglobin A1c (HbA1c) ≤7.5 % based on central laboratory screening results.
* Fasting C-peptide <0.6 nanograms per milliliter (ng/mL).
* Participants should be in good general health based on medical history and physical examination and without medical conditions that might prevent the completion of study drug injections and assessments required in this protocol.

Exclusion Criteria:

* Known or suspected allergy to any component of any of the study drugs in this study.
* Previous enrollment in this study. Participants who fail Screening may attempt to rescreen into the study.
* A participant who has proliferative retinopathy or maculopathy, and/or severe neuropathy, in particular autonomic neuropathy, as judged by the Investigator.
* As judged by the Investigator, clinically significant active disease of the gastrointestinal, cardiovascular (including a history of arrhythmia or conduction delays on electrocardiogram [ECG]), hepatic, neurological, renal, genitourinary, or hematological systems.
* As judged by the Investigator, uncontrolled hypertension (diastolic blood pressure ≥100 millimeters of mercury [mmHg] and/or systolic blood pressure ≥160 mmHg after 5 minutes in the supine position). Three attempts may be performed to measure blood pressure.
* History of any illness or disease that in the opinion of the Investigator might confound the results of the study or pose additional risk in administering the study drugs to the participant.
* As judged by the Investigator, clinically significant findings in routine laboratory data.
* Use of drugs (such as systemic corticosteroids) that may interfere with the interpretation of study results or are known to cause clinically relevant interference with insulin action, glucose utilization, or recovery from hypoglycemia.
* Recurrent severe hypoglycemia (more than 2 episodes over the last 6 months) or hypoglycemic unawareness, as judged by the Investigator.
* Current addiction to alcohol or substances of abuse, as determined by the Investigator.
* Pregnancy, breast-feeding, the intention of becoming pregnant, or not using adequate contraceptive measures (adequate contraceptive measures consist of sterilization, intra-uterine device [IUD], oral or injectable contraceptives, or barrier methods).
* Mental incapacity, unwillingness, or language barriers precluding adequate understanding or cooperation in this study.
* Receipt of any investigational drug within 4 weeks of Screening.
* Any condition (intrinsic or extrinsic) that in the judgment of the Investigator will interfere with study participation or evaluation of data. Examples would include: renal insufficiency (serum creatinine >1.5 milligrams per deciliter [mg/dL] for males or >1.4 mg/dL for females), congestive heart failure required medication treatment, and cardiac disease with New York Heart Association (NYHA) Functional Capacity of III/IV.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2009-05; Primary Completion 2010-02 (Actual); Study Completion 2010-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Douglas Muchmore, M.D., Study Director — Halozyme Therapeutics
Locations (8):
- United States (8):
  - Barbara Davis Center for Childhood Diabetes, Aurora, Colorado
  - Diabetes Research Institute, Miami, Florida
  - Henry Ford Health System, Detroit, Michigan
  - Mercury Street Medical, Butte, Montana
  - UNC Diabetes Care Center/Highgate Specialty Center, Durham, North Carolina
  - Cleveland Clinic, Cleveland, Ohio
  - Texas Diabetes and Endocrinology, Austin, Texas
  - West Olympia Internal Medicine, Olympia, Washington

RESULTS

PARTICIPANT FLOW:
Groups:
- All Enrolled Participants: Prior to randomization, all enrolled participants underwent a 1-month dose titration period.
  Insulin Lispro (Titration Period): 100 units per milliliter (U/mL), injected subcutaneously before meals, with doses titrated to each individual participant's glycemic control needs, for 1 month.
  Participants requiring basal insulin used twice daily, subcutaneous injections of 100 U/mL insulin glargine or maintained their usual regimen through an infusion pump.
- INSULIN-PH20 NP First, Then Insulin Lispro: Following a 1-month dose titration period, participants were randomly assigned to Treatment A for the first 3-month treatment cycle, followed by Treatment B for the second 3-month treatment cycle.
  INSULIN-PH20 NP (Treatment A): 100 units per milliliter (U/mL) non-preserved (NP) formulation of recombinant human insulin with 5.0 micrograms per milliliter (µg/mL) recombinant human hyaluronidase PH20, injected subcutaneously before meals, with doses titrated to each individual participant's glycemic control needs, for 3 months.
  Insulin Lispro (Treatment B): 100 U/mL insulin lispro, injected subcutaneously before meals, with doses titrated to each individual participant's glycemic control needs, for 3 months.
  Participants requiring basal insulin used twice daily, subcutaneous injections of 100 U/mL insulin glargine or maintained their usual regimen through an infusion pump.
- Insulin Lispro First, Then INSULIN-PH20 NP: Following a 1-month dose titration period, participants were randomly assigned to Treatment B for the first 3-month treatment cycle, followed by Treatment A for the second 3-month treatment cycle.
  Insulin Lispro (Treatment B): 100 units per milliliter (U/mL) insulin lispro, injected subcutaneously before meals, with doses titrated to each individual participant's glycemic control needs, for 3 months.
  INSULIN-PH20 NP (Treatment A): 100 U/mL non-preserved (NP) formulation of recombinant human insulin with 5.0 micrograms per milliliter (µg/mL) recombinant human hyaluronidase PH20, injected subcutaneously before meals, with doses titrated to each individual participant's glycemic control needs, for 3 months.
  Participants requiring basal insulin used twice daily, subcutaneous injections of 100 U/mL insulin glargine or maintained their usual regimen through an infusion pump.
Period: Titration Period (Weeks 0 to 4)
Arm/Group | All Enrolled Participants | INSULIN-PH20 NP First, Then Insulin Lispro | Insulin Lispro First, Then INSULIN-PH20 NP
Started | 48 | 0 | 0
Completed | 46 | 0 | 0
Not Completed | 2 | 0 | 0
Not completed — Withdrawal by Subject | 2 | 0 | 0
Period: First Treatment Cycle (Weeks 4 to 16)
Arm/Group | All Enrolled Participants | INSULIN-PH20 NP First, Then Insulin Lispro | Insulin Lispro First, Then INSULIN-PH20 NP
Started | 0 | 22 | 24
Received at Least 1 Dose of Study Drug | 0 | 22 | 24
Completed | 0 | 19 | 23
Not Completed | 0 | 3 | 1
Not completed — Adverse Event | 0 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 1
Not completed — Protocol Violation | 0 | 1 | 0
Period: Second Treatment Cycle (Weeks 16 to 28)
Arm/Group | All Enrolled Participants | INSULIN-PH20 NP First, Then Insulin Lispro | Insulin Lispro First, Then INSULIN-PH20 NP
Started | 0 | 19 | 23
Received at Least 1 Dose of Study Drug | 0 | 19 | 23
Completed | 0 | 19 | 22
Not Completed | 0 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Participants who were randomized and received at least 1 dose of study drug.
Groups:
- All Randomized Participants: Following a 1-month titration period, participants were randomly assigned to 1 of 2 study treatments (Treatment A or B) for the first of two, 3-month treatment cycles. Each participant then received the second treatment for the second cycle.
  INSULIN-PH20 NP (Treatment A): 100 U/mL non-preserved (NP) formulation of regular human insulin with 5.0 micrograms per milliliter (µg/mL) recombinant human hyaluronidase PH20, injected SC, pre-meals, doses titrated to each participant individually.
  Insulin Lispro (Treatment B): 100 U/mL insulin lispro, injected SC, pre-meals, doses titrated to each participant individually.
  Throughout the study, participants requiring basal insulin used twice daily SC injections of 100 U/mL insulin glargine or maintained their usual regimen through an insulin pump.
Arm/Group | All Randomized Participants
Number analyzed (Participants) | 46
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.6 (13.28)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22
  Male | 24
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 44
  More than one race | 0
  Unknown or Not Reported | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 44
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 46

OUTCOME MEASURES:

1. Primary Outcome: Postprandial Glucose Excursion
Description: A 2-hour postprandial glucose excursion was measured for 3 meals over 3 days during each treatment cycle (3 days during Week 14 of the first treatment cycle and 3 days during Week 26 of the second treatment cycle). For each of the 3 days, the mealtime (breakfast, lunch, and dinner) excursions were calculated as the post-meal glucose value minus the pre-meal value as determined by 8-point glucose monitoring. The average of all excursions over the 3 days for the corresponding treatment cycle is presented.
Time Frame: Week 14 and Week 26
Population: Participants who completed both treatment cycles with evaluable postprandial glucose data.
Measure: Mean (Standard Deviation); unit: milligrams per deciliter (mg/dL)
Groups:
- INSULIN-PH20 NP: 100 units per milliliter (U/mL) non-preserved formulation of recombinant human insulin with 5.0 micrograms per milliliter (µg/mL) recombinant human hyaluronidase (INSULIN-PH20 NP), injected subcutaneously before meals, with doses titrated to each individual participant's glycemic control needs, for 3 months.
- Insulin Lispro: 100 units per milliliter (U/mL) insulin lispro, injected subcutaneously before meals, with doses titrated to each individual participant's glycemic control needs, for 3 months.
Arm/Group | INSULIN-PH20 NP | Insulin Lispro
Number analyzed (Participants) | 37 | 37
milligrams per deciliter (mg/dL) | 17.23 (36.040) | 14.47 (35.113)
Statistical Analysis 1: Comparison: INSULIN-PH20 NP vs Insulin Lispro; A total of at least 40 participants were to be enrolled in the study, and 30 participants were expected to complete both treatment cycles. Assuming a standard deviation for blood glucose of 45 milligrams per deciliter (mg/dL) and a true difference between the treatments of 0 mg/dL, the study had approximately 80% power to show that INSULIN-PH20 NP was non-inferior to insulin lispro with respect to the overall two-hour postprandial blood glucose excursion; Test type: Non-Inferiority or Equivalence — Non-inferiority of INSULIN-PH20 NP to insulin lispro was supported if the upper limit of the one-sided 95% confidence interval for the difference in blood glucose between the treatments did not exceed 21.6 mg/dL; p = 0.3217, Mixed Models Analysis; Adjustments included treatment, phase, and treatment sequence as fixed effects and participant within treatment sequence as a random effect; LS Mean Difference = 3.06, 95% CI 1-sided [upper limit 14.11]

2. Secondary Outcome: Time Spent With Blood Glucose Value Outside a 71-139 Milligrams Per Deciliter (mg/dL) Range During Continuous Glucose Monitoring
Description: Participants were provided a continuous glucose monitoring (CGM) device, consisting of a sensor, transmitter, and receiver. Total time the participant's blood glucose was outside the 71-139 mg/dL range during 3 days of CGM during each treatment cycle (3 days during Week 14 of the first treatment cycle and 3 days during Week 26 of the second treatment cycle) is presented.
Time Frame: Week 14 and Week 26
Population: Participants that completed both treatment cycles with evaluable CGM data.
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | INSULIN-PH20 NP | Insulin Lispro
Number analyzed (Participants) | 40 | 40
hours | 14.58 (3.155) | 13.37 (3.933)

3. Secondary Outcome: Number of Participants With Hypoglycemic Events
Description: The number of participants with at least one hypoglycemic event (HE) reported during the entire study is presented. Additionally, the number of participants with severe HEs (those that necessitated administration of carbohydrate or glucagon, or resuscitation, by another person) is also presented. A summary of serious and other non-serious adverse events regardless of causality is located in the Reported Adverse Events module.
Time Frame: Baseline through Week 29
Population: Participants who received at least 1 dose of study drug.
Measure: Number; unit: participants
Arm/Group | INSULIN-PH20 NP | Insulin Lispro
Number analyzed (Participants) | 45 | 43
participants
  Overall | 45 | 43
  Severe HE | 2 | 0

ADVERSE EVENTS:
Time Frame: An adverse event was considered treatment-emergent if the start date of the event was on or after the date of randomization.
Groups:
- INSULIN-PH20 NP Treatment Period: 100 units per milliliter (U/mL) non-preserved formulation of recombinant human insulin with 5.0 micrograms per milliliter (µg/mL) recombinant human hyaluronidase (INSULIN-PH20 NP), injected subcutaneously before meals, with doses titrated to each individual participant's glycemic control needs, for 3 months.
- Insulin Lispro Treatment Period: 100 units per milliliter (U/mL) insulin lispro, injected subcutaneously before meals, with doses titrated to each individual participant's glycemic control needs, for 3 months.
Arm/Group | INSULIN-PH20 NP Treatment Period | Insulin Lispro Treatment Period
Serious Adverse Events (participants affected / at risk) | 2/45 | 1/43
Other Adverse Events (participants affected / at risk) | 17/45 | 11/43
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | INSULIN-PH20 NP Treatment Period (N=45) | Insulin Lispro Treatment Period (N=43)
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Uterine haemorrhage (Reproductive system and breast disorders) | 1/22 (1) | 0/20 (0)
Haemothorax (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Rib fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | INSULIN-PH20 NP Treatment Period (N=45) | Insulin Lispro Treatment Period (N=43)
Nasopharyngitis (Infections and infestations) | 7 (7) | 7 (8)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 3 (3)
Sinusitis (Infections and infestations) | 2 (2) | 1 (1)
Bronchitis (Infections and infestations) | 2 (2) | 0 (0)
Fungal infection (Infections and infestations) | 2 (2) | 1 (1)
Food poisoning (Gastrointestinal disorders) | 0 (0) | 2 (2)
Injection site haematoma (General disorders) | 2 (3) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Hypoglycaemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Hypertension (Vascular disorders) | 2 (2) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
All information obtained as a result of this study or during the conduct of this study will be regarded as confidential. The investigator agrees to use the information for the purpose of carrying out this study and for no other purpose, unless written permission from the sponsor (Halozyme) is obtained.